CLINICAL TRIAL: NCT07049211
Title: Individualized Closed-Loop Neuromodulation With Repetitive Transcranial Magnetic Stimulation Synchronized Task Training for Upper Limb Motor Dysfunction in Stroke Patients
Brief Title: Individualized rTMS Synchronized Task Training for Closed-loop Neuromodulation of Post-stroke Motor Dysfunction
Acronym: rTMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: shanghai center for brain science and brain-inspired technology (Unknown)
Responsible Party: Principal Investigator, Qing Xie, PhD, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025296
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Upper Extremity Dysfunction After the Stroke
Keywords: repetitive transcranial magnetic stimulaiton; stroke; online; individualized; upper limb motor dysfunction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized online stimulation (Experimental): The individualized online stimulation group will calculate precise targets based on the collected multimodal MRI (structural images, resting-state/task-state functional images, and diffusion tensor imaging), plan the coil position and placement angle of TMS through electric field simulation, and achieve individualized intervention. At the same time, when patients receive TMS treatment, they are paired with specific upper limb motor tasks. When the task starts autonomously, TMS stimulation is triggered by acceleration-EMG feedback. When the task stops or is completed, TMS stimulation also stops immediately according to the acceleration-EMG feedback to achieve real-time effects.
  Interventions: Device: Individualized online stimulation
- Non-individualized online stimulation (Active Comparator): In the non-individualized online stimulation group, patients receive TMS treatment synchronized with task training. However, the targeting uses traditional positioning methods, i.e., determining the target with a positioning cap instead of precise target localization.
  Interventions: Device: Non-individualized online stimulation
- Sham stimulation (Sham Comparator): In the individualized online sham stimulation group, patients receive TMS treatment combined with specific tasks. The stimulation targets are the same as those in the online stimulation group, all determined by precise target localization, except that a sham stimulation coil is used for TMS stimulation.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Individualized online stimulation — The individualized online stimulation group will calculate precise targets based on the collected multimodal MRI (structural images, resting-state/task-state functional images, and diffusion tensor imaging), plan the coil position and placement angle of TMS through electric field simulation, and achieve individualized intervention. At the same time, when patients receive TMS treatment, they are matched with specific upper limb motor tasks. When the task starts autonomously, TMS stimulation is triggered by acceleration-EMG feedback. When the task stops or is completed, TMS stimulation also stops immediately according to the acceleration-EMG feedback to achieve real-time effects.
  Arms: Individualized online stimulation
Device: Non-individualized online stimulation — In the non-individualized online stimulation group, patients receive TMS treatment synchronized with task training. However, the targeting uses traditional positioning methods, i.e., determining the target with a positioning cap instead of precise target localization.
  Arms: Non-individualized online stimulation
Device: Sham stimulation — In the individualized online sham stimulation group, patients receive TMS treatment combined with specific tasks. The stimulation targets are the same as those in the online stimulation group, all determined by precise target localization, except that a sham stimulation coil is used for TMS stimulation.
  Arms: Sham stimulation

SUMMARY:
The goal of this clinical trials is to investigate the effectiveness of individualized online repetitive transcranial magnetic stimulation (rTMS) in enhancing upper limb motor rehabilitation during the subacute and chronic phase of stroke. It will also learn about the safety of online rTMS intervention methods. The main questions it aims to answer are:

1. Does individualized rTMS precise target combined with motor training improve upper limb motor rehabilitation in patients？
2. Does individualized rTMS precise target combined with motor training enhance the upper limb motor rehabilitation ability in stroke patients by strengthening the functional coupling of the motor circuit to achieve functional reorganization of the brain network ?

Researchers will compare individualized online rTMS to non-individualized online and individualized sham stimulation in stroke patients to see if individualized online rTMS works to alleviate motor dysfunction in this randomized，sham-controlled, double-blind trial.

Participants will:

1. randomized to one group(individualized online, non-individualized online or sham);
2. receive rTMS treatment for 10 days, with 5 working days per week for a total of two weeks;
3. receive magnetic resonance imaging (MRI) and electroencephalogram (EEG) evaluations before and after the entire treatment;
4. conduct scales and MEP assessment one day before the treatment, as well as one day, one month, and three months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is first diagnosed with stroke through neurological examination, CT or MRI scan.
2. The vital signs are stable and there is a certain degree of upper limb motor dysfunction.
3. Motor evoked potentials(MEPs) of First Dorsal Interosseous Muscle（FDI）or Abductor Pollicis Brevis Muscle (APB) is negative in ipsilesional hemisphere.
4. The age is between 20 and 80 years old.
5. The cognitive ability is not significantly affected and the patient can cooperate with various examinations and assessments, with a MMSE score ≥ 20 points.
6. There are no serious complications (such as pneumonia, heart failure, urinary tract infection or malnutrition).
7. There is no pathological condition that is a contraindication for TMS in the medical history (for example, patients with metal in the brain, such as aneurysm clips, patients with a cardiac pacemaker, pregnant women, or those with a history of epileptic seizures).
8. The patient or guardian agrees to sign the informed consent form.

Exclusion Criteria:

1. Patients with severe heart, lung, liver, kidney diseases and malignant tumors;
2. Those with a history of aphasia, severe cognitive impairment or mental illness;
3. Patients who have had a history of epileptic seizures in the last month or are taking anti-epileptic drugs recently;
4. Those with severe visual or hearing impairments, unable to communicate normally;
5. People with metal implants, pacemakers, skull defects or other conditions that prevent them from undergoing TMS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity (FMA-UE) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 90 after 2-week intervention
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The Fugl-Meyer Assessment - Upper Extremity (FMA-UE) is the upper limb motor domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, hand. It ranges from 0 (hemiplegia) to 66 points (normal motor performance).

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 90 after 2-week intervention
  The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery, brain injury and multiple sclerosis populations. The ARAT was originally described by Lyle in 1981 as a modified version of the Upper Extremity Function Test and was used to examine upper limb functional recovery post damage to the cortex.
Modified Barthel Index (MBI) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 90 after 2-week intervention
  The Barthel Index for activities of daily living was introduced in 1965 by Barthel and Mahoney to be used in the assessment of the degree of assistance required by patients with stroke (other neuromuscular or musculoskeletal disorders or oncology patients) with regards to 10 items of mobility and self-care (ADL).
The Pittsburgh Sleep Quality Index (PSQI) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 90 after 2-week intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. The PSQI is commonly used in both clinical and research settings to evaluate various aspects of sleep. It is a valuable tool for assessing sleep quality as it captures multiple dimensions of sleep, including both subjective experiences and objective parameters. It allows researchers and healthcare providers alike to obtain a comprehensive understanding of an individual's sleep patterns and disturbances and inform treatment decisions and interventions for sleep disorders.
Motor Evoked Potential (MEP) - Resting Motor Threshold (RMT) | Baseline; Day 6 during 2-week intervention; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 90 after 2-week intervention
  Resting motor threshold is an objective measure of cortical excitability. Numerous studies indicate that the success of motor recovery after stroke is significantly determined by the direction and extent of cortical excitability changes.
The average completion time for baseline tasks | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day7, Day 8, Day 9, Day 10 during TMS intervention
  The average completion time for baseline tasks refers to the time (seconds) taken by the patient to complete the baseline motor task before each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Wang, PhD, Study Director — shanghai center for brain science and brain-inspired technology
Locations (1):
- Shanghai Ruijin Hospital, affiliated to Shanghai Jiao Tong University, School of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will share the demographic information and baseline clinical data of all participants.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Authorized professional researchers, including but not limited to researchers engaged in neuroscience research who have obtained data access permission from their affiliated institutions, and clinical doctors from other medical institutions that have a cooperative relationship with this study and have signed data confidentiality agreements.
  They can access the detailed clinical medical histories of the participants, including past disease histories and treatment process records; neurological function assessment scale data; as well as imaging data collected during the study, such as brain magnetic resonance imaging (MRI) results. However, sensitive information related to participants' privacy, such as names, ID numbers, and contact information, will be strictly anonymized to ensure that such information cannot be obtained.
  They can contact the corresponding author or the first author via email.
URL: https://zenodo.org/records/15672312

REFERENCES:
- [Background] Khedr EM, Etraby AE, Hemeda M, Nasef AM, Razek AA. Long-term effect of repetitive transcranial magnetic stimulation on motor function recovery after acute ischemic stroke. Acta Neurol Scand. 2010 Jan;121(1):30-7. doi: 10.1111/j.1600-0404.2009.01195.x. Epub 2009 Aug 11. PMID 19678808
- [Background] Ackerley SJ, Stinear CM, Barber PA, Byblow WD. Combining theta burst stimulation with training after subcortical stroke. Stroke. 2010 Jul;41(7):1568-72. doi: 10.1161/STROKEAHA.110.583278. Epub 2010 May 20. PMID 20489170
- [Background] Xiang H, Sun J, Tang X, Zeng K, Wu X. The effect and optimal parameters of repetitive transcranial magnetic stimulation on motor recovery in stroke patients: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2019 May;33(5):847-864. doi: 10.1177/0269215519829897. Epub 2019 Feb 18. PMID 30773896
- [Background] Zhang L, Xing G, Fan Y, Guo Z, Chen H, Mu Q. Short- and Long-term Effects of Repetitive Transcranial Magnetic Stimulation on Upper Limb Motor Function after Stroke: a Systematic Review and Meta-Analysis. Clin Rehabil. 2017 Sep;31(9):1137-1153. doi: 10.1177/0269215517692386. Epub 2017 Feb 17. PMID 28786336
- [Background] van Lieshout ECC, van der Worp HB, Visser-Meily JMA, Dijkhuizen RM. Timing of Repetitive Transcranial Magnetic Stimulation Onset for Upper Limb Function After Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2019 Dec 3;10:1269. doi: 10.3389/fneur.2019.01269. eCollection 2019. PMID 31849827
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Kim JH. Effects of a virtual reality video game exercise program on upper extremity function and daily living activities in stroke patients. J Phys Ther Sci. 2018 Dec;30(12):1408-1411. doi: 10.1589/jpts.30.1408. Epub 2018 Nov 21. PMID 30568325
- [Background] Diekhoff-Krebs S, Pool EM, Sarfeld AS, Rehme AK, Eickhoff SB, Fink GR, Grefkes C. Interindividual differences in motor network connectivity and behavioral response to iTBS in stroke patients. Neuroimage Clin. 2017 Jun 4;15:559-571. doi: 10.1016/j.nicl.2017.06.006. eCollection 2017. PMID 28652969
- [Background] Li CT, Huang YZ, Bai YM, Tsai SJ, Su TP, Cheng CM. Critical role of glutamatergic and GABAergic neurotransmission in the central mechanisms of theta-burst stimulation. Hum Brain Mapp. 2019 Apr 15;40(6):2001-2009. doi: 10.1002/hbm.24485. Epub 2019 Jan 1. PMID 30600571
- [Background] Zhang L, Xing G, Shuai S, Guo Z, Chen H, McClure MA, Chen X, Mu Q. Low-Frequency Repetitive Transcranial Magnetic Stimulation for Stroke-Induced Upper Limb Motor Deficit: A Meta-Analysis. Neural Plast. 2017;2017:2758097. doi: 10.1155/2017/2758097. Epub 2017 Dec 21. PMID 29435371
- [Background] Dionisio A, Duarte IC, Patricio M, Castelo-Branco M. The Use of Repetitive Transcranial Magnetic Stimulation for Stroke Rehabilitation: A Systematic Review. J Stroke Cerebrovasc Dis. 2018 Jan;27(1):1-31. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.008. Epub 2017 Oct 27. PMID 29111342
- [Background] Graef P, Dadalt MLR, Rodrigues DAMDS, Stein C, Pagnussat AS. Transcranial magnetic stimulation combined with upper-limb training for improving function after stroke: A systematic review and meta-analysis. J Neurol Sci. 2016 Oct 15;369:149-158. doi: 10.1016/j.jns.2016.08.016. Epub 2016 Aug 12. PMID 27653882
- [Background] Houdayer E, Degardin A, Cassim F, Bocquillon P, Derambure P, Devanne H. The effects of low- and high-frequency repetitive TMS on the input/output properties of the human corticospinal pathway. Exp Brain Res. 2008 May;187(2):207-17. doi: 10.1007/s00221-008-1294-z. Epub 2008 Feb 8. PMID 18259738
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Lin YL, Potter-Baker KA, Cunningham DA, Li M, Sankarasubramanian V, Lee J, Jones S, Sakaie K, Wang X, Machado AG, Plow EB. Stratifying chronic stroke patients based on the influence of contralesional motor cortices: An inter-hemispheric inhibition study. Clin Neurophysiol. 2020 Oct;131(10):2516-2525. doi: 10.1016/j.clinph.2020.06.016. Epub 2020 Jul 3. PMID 32712080
- [Background] Cicinelli P, Pasqualetti P, Zaccagnini M, Traversa R, Oliveri M, Rossini PM. Interhemispheric asymmetries of motor cortex excitability in the postacute stroke stage: a paired-pulse transcranial magnetic stimulation study. Stroke. 2003 Nov;34(11):2653-8. doi: 10.1161/01.STR.0000092122.96722.72. Epub 2003 Oct 9. PMID 14551397
- [Background] Murase N, Duque J, Mazzocchio R, Cohen LG. Influence of interhemispheric interactions on motor function in chronic stroke. Ann Neurol. 2004 Mar;55(3):400-9. doi: 10.1002/ana.10848. PMID 14991818
- [Background] Nowak DA, Grefkes C, Ameli M, Fink GR. Interhemispheric competition after stroke: brain stimulation to enhance recovery of function of the affected hand. Neurorehabil Neural Repair. 2009 Sep;23(7):641-56. doi: 10.1177/1545968309336661. Epub 2009 Jun 16. PMID 19531606
- [Background] Ridding MC, Rothwell JC. Is there a future for therapeutic use of transcranial magnetic stimulation? Nat Rev Neurosci. 2007 Jul;8(7):559-67. doi: 10.1038/nrn2169. PMID 17565358
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Hachinski V, Donnan GA, Gorelick PB, Hacke W, Cramer SC, Kaste M, Fisher M, Brainin M, Buchan AM, Lo EH, Skolnick BE, Furie KL, Hankey GJ, Kivipelto M, Morris J, Rothwell PM, Sacco RL, Smith SC Jr, Wang Y, Bryer A, Ford GA, Iadecola C, Martins SC, Saver J, Skvortsova V, Bayley M, Bednar MM, Duncan P, Enney L, Finklestein S, Jones TA, Kalra L, Kleim J, Nitkin R, Teasell R, Weiller C, Desai B, Goldberg MP, Heiss WD, Saarelma O, Schwamm LH, Shinohara Y, Trivedi B, Wahlgren N, Wong LK, Hakim A, Norrving B, Prudhomme S, Bornstein NM, Davis SM, Goldstein LB, Leys D, Tuomilehto J. Stroke: working toward a prioritized world agenda. Int J Stroke. 2010 Aug;5(4):238-56. doi: 10.1111/j.1747-4949.2010.00442.x. PMID 20636706
- [Background] Dionisio A, Duarte IC, Patricio M, Castelo-Branco M. Transcranial Magnetic Stimulation as an Intervention Tool to Recover from Language, Swallowing and Attentional Deficits after Stroke: A Systematic Review. Cerebrovasc Dis. 2018;46(3-4):178-185. doi: 10.1159/000494213. Epub 2018 Oct 19. PMID 30343304
- [Background] Feigin VL, Barker-Collo S, Parag V, Senior H, Lawes CM, Ratnasabapathy Y, Glen E; ASTRO study group. Auckland Stroke Outcomes Study. Part 1: Gender, stroke types, ethnicity, and functional outcomes 5 years poststroke. Neurology. 2010 Nov 2;75(18):1597-607. doi: 10.1212/WNL.0b013e3181fb44b3. PMID 21041783
- [Background] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Background] Feigin VL, Lawes CM, Bennett DA, Barker-Collo SL, Parag V. Worldwide stroke incidence and early case fatality reported in 56 population-based studies: a systematic review. Lancet Neurol. 2009 Apr;8(4):355-69. doi: 10.1016/S1474-4422(09)70025-0. Epub 2009 Feb 21. PMID 19233729
- [Background] Hatano S. Experience from a multicentre stroke register: a preliminary report. Bull World Health Organ. 1976;54(5):541-53. PMID 1088404
- See also: The URL is the data sharing website of this study, which briefly describes the protocol and objectives of the research. — https://zenodo.org/records/15672312
- Available data/document: Individual Participant Data Set — https://zenodo.org/records/15672312 — Method of obtaining the raw data: If there are reasonable requests, the related raw data to support the research results can be obtained from the corresponding authors or the first authors. Data sharing website: https://zenodo.org/records/15080604 Time of making the raw data public: the research raw data will be publicly shared six months after the publication of the research paper.
- Available data/document: Study Protocol — https://zenodo.org/records/15672312 — Method of obtaining the raw data: If there are reasonable requests, the related raw data to support the research results can be obtained from the corresponding authors or the first authors. Data sharing website: https://zenodo.org/records/15080604 Time of making the raw data public: the research raw data will be publicly shared six months after the publication of the research paper.
- Available data/document: Analytic Code — https://zenodo.org/records/15672312 — Method of obtaining the raw data: If there are reasonable requests, the related raw data to support the research results can be obtained from the corresponding authors or the first authors. Data sharing website: https://zenodo.org/records/15080604 Time of making the raw data public: the research raw data will be publicly shared six months after the publication of the research paper.